CLINICAL TRIAL: NCT04518020
Title: Single Crown Supported by Short Implant Versus Standard Implant in Conjunction With Maxillary Sinus Floor Augmentation in the Posterior: a Randomized, Controlled Clinical Trial.
Brief Title: Single Crown Supported by Short Implant Versus Standard Implant in Conjunction With Maxillary Sinus Floor Augmentation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Principal Investigator, Helle Baungaard Nielsen, Principal Investigator, PhD. Student, Department of Oral and Maxillofacial Surgery, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20160047
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short implant (Active Comparator): Short implant 6 mm installed
  Interventions: Procedure: 40 patients will be randomly allocated to short implants and standard implants in conjunction with MSFA
- Conventional implant + bone augmentation (Other): Standard length implant 13 mm in conjunction with maxillary sinus floor augmentation serves as a control group
  Interventions: Procedure: 40 patients will be randomly allocated to short implants and standard implants in conjunction with MSFA

INTERVENTIONS:
Procedure: 40 patients will be randomly allocated to short implants and standard implants in conjunction with MSFA — 40 patients will be randomly allocated to short implants (group 1) and standard implants in conjunction with MSFA using 50% particulated autogenous mandibular bone graft mixed with 50% Bio-Oss (group 2).

SUMMARY:
Implant placement in the posterior part of the maxilla is frequently compromised due to atrophy of the alveolar process. Therefore, alveolar ridge augmentation is frequently necessary before or in conjunction with implant placement. The most commonly used method to augment the maxillary premolar and molar region involves the maxillary sinus floor augmentation (MSFA) with autogenous bone graft or a bone substitute. However, the use of autogenous bone grafts is associated with risk at the donor site morbidity and unpredictable graft resorption. Consequently, short implants are used increasingly to eliminate the need for bone augmentation. However, long-term studies comparing short implants and standard implants in conjunction with MSFA supporting single crown restoration in the posterior maxilla are missing. The primary outcome measures include survival of implant and suprastructures, peri-implant marginal bone level (MBL), professional evaluation of the suprastructure and soft tissue using pink esthetic score (PES) and white esthetic score (WES), patient satisfaction using visual analogue scale (VAS), and oral health related quality of life using oral health impact profile (OHIP-14) questionnaire. Secondary outcome measure include evaluation of the complication rate related to the two treatment modalities.

DETAILED DESCRIPTION:
The primary objective of the present study is to test the H0 hypothesis of:

1. No differences in survival of suprastructures and implants with the two treatment modalities.
2. No differences in peri-implant MBL, PES, WES, and patient satisfaction using VAS with the two treat modalities.
3. No differences in oral health related quality of life using OHIP-14 with the two treatment modalities.

The secondary objective will include:

1. Complications related to bone harvesting, implant installation, and MSFA.

The primary outcome measures included:

* Survival of suprastructures.
* Survival of implants.
* Radiographic peri-implant MBL.
* Professional evaluation of suprastructure and soft tissue using PES and WES.
* Patient satisfaction using VAS
* Oral health related quality of life using OHIP-14 questionnaire.

Secondary outcome measures:

• Pre- and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* >20 years
* Partial edentulism in the posterior maxilla.
* Height and weight of the maxillary alveolar process of at least 5.5 mm.
* Mandibular occluding teeth.

Exclusion Criteria:

* General contraindications to implant therapy.
* Poor oral hygiene.
* Progressive periodontitis.
* Acute infection in the area intended for implant placement.
* Parafunction, bruxism, or clenching.
* Psychiatric problems or unrealistic expectations.
* Heavy tobacco use, define as >10 cigarettes per day.
* Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Survival of suprastructures. | 1-year follow up
  Survival of suprastructures is defined as absence of mechanical/or biological complications causing loss of suprastructures. Chipping of ceramics and loosening of the suprastructure were not categorized as loss of suprastructure.
Survival of implants. | 1-year follow up
  Survival of implants is defined as clinically stable and osseointegrated implants with absence of mobility, progressive marginal bone loss, and infection.
Radiographic MBL. | 1-year follow up
  Measurement of marginal bone level in millimeter.
Professional evaluation of the prosthetic restoration and soft tissue using pink esthetic score (PES) and white esthetic score (WES). | 1-year follow up
  Esthetic evaluation of suprastructure and soft tissue using PES and WES. PES includes 7 different variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue colour, and texture. Each variable is assessed with a 0, 1, or 2 score, with 0 being the poorest score and 2 the best according to the degree of match or mismatch compared with the anterior premolar or molar. The highest possible PES is 14. WES includes 5 different variables: Crown form, volume, colour, translucency, and texture. Each variable is assessed with a 0, 1, or 2 score, with 0 being the poorest score and 2 the best according to the degree of match or mismatch compared with the anterior premolar or molar. The highest possible WES is 10.
Patient satisfaction. | 1-year follow up
  Evaluation of patient satisfaction using visual analogue scale (VAS). VAS with 0 indicating extreme dissatisfaction and 10 indicating complete satisfaction.
Oral health related quality of life as defined by oral health impact profile (OHIP-14). | 1-year follow up
  Evaluation of oral health related quality of life using OHIP-14 questionnaire. OHIP-14 scale ranges from 0 to 56, with higher scores indicating poorer oral health impact profile.

SECONDARY OUTCOMES:
Complications. | 1-year follow up
  Evaluation of biological and mechanical complication rate.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nielsen HB, Schou S, Bruun NH, Starch-Jensen T. Single-crown restorations supported by short implants (6 mm) compared with standard-length implants (13 mm) in conjunction with maxillary sinus floor augmentation: a randomized, controlled clinical trial. Int J Implant Dent. 2021 Jul 16;7(1):66. doi: 10.1186/s40729-021-00348-5. PMID 34268630